CLINICAL TRIAL: NCT06220695
Title: Efficacy of Isocaloric Mediterranean Diet and Low-fat Diet in Overweight/Obese MASLD Subjects With Respect to PNPLA3 Single Nucleotide Polymorphism: A Randomized Controlled Trial
Brief Title: A Nutrigenetic Intervention in MASLD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMCRPS-23-1
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: NAFLD; Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet Group (Experimental): The Mediterranean diet includes high amounts of olive oil, olives, fruits, vegetables, whole grains, legumes, nuts, a high intake of fish, moderate consumption of eggs, poultry, and dairy, and low consumption of red meat and products. The targeted macronutrient distribution is 40% of total energy from carbohydrates, approximately 20% from protein, and 40% from fats. The share of saturated fats in total energy will not exceed 10%. Participants will be provided with written resources, brochures explaining the Mediterranean diet, and information about the Mediterranean diet pyramid. A weekly menu will be planned for all participants, along with cooking tips.
  Participants in this group will receive a weekly food support package for 12 weeks, including essential elements of the Mediterranean diet such as olive oil, fish, nuts, and legumes.
  Interventions: Behavioral: Dietary intervention
- Low Fat Diet Group (Active Comparator): The type of diet to be followed in this group is based on the recommendations of the American Heart Association, the American Diabetes Association guidelines, and the Specific Nutrition Guide for Turkey. The targeted macronutrient distribution will be 50% of total energy from carbohydrates, approximately 20% from protein, and less than 30% from fats. The share of saturated fats in total energy will not exceed 10%. Participants will be provided with information notes and brochures explaining the low-fat diet. A weekly menu will be planned for all participants, and cooking tips will be provided.
  Participants in this group will receive a weekly food support package for 12 weeks, including low-fat dairy products, whole grains, and legumes, which are the essential elements of a low-fat diet.
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — The dietary intervention is a personalized counselling programme implemented in form of a moderate caloric restriction (≈500 kcal/day) to allow for a moderate weight loss (≈5% BW). Each participant will be invited for consultation visits to a study dietitian, lasting up to 30 minutes. During the sessions, participants will be provided with written information material that explains the principles of diet in concern. Dietary interventions for both groups will be standardized in terms of education and one-on-one counseling. Education and dietary prescription will be individualized by the study dietitians within the diet-specific recommendations, to allow for personal food preferences. All subjects will receive equivalent intensity of care in terms of opportunities for contact and availability of individual dietary counseling. Motivational interviewing techniques and behavior change techniques will be adopted by study dietitians to ensure long-term maintenance of dietary modification.

SUMMARY:
The study is designed as a 12-week randomized controlled dietary intervention in individuals who had been diagnosed with NAFLD in the last 6 months and whose body mass index is above 25 at the time of participation in the pre-screening. The study sample is determined as 150 subjects and randomization will be done by stratification according to PNPLA3 genotype. At baseline, hepatic steatosis and fibrosis will be measured with Fibroscan, body composition will be analyzed, and transaminases and sugar and lipid metabolism indicators will be examined. The study will be conducted in parallel groups, with each group receiving equal amounts and intensity of Mediterranean diet or low-fat diet therapy. At the end of the 12-week intervention, baseline measurements will be repeated and the efficacy of the Mediterranean Diet and Low-fat diet therapies will be compared, as well as the effect of PNPLA3 mutation on intrahepatic response will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign informed consent
* BMI> 25 kg/m2
* Between 18-80 years
* previous clinical diagnosis of MASLD by abdominal USG, MRI, FibroScan® or liver biopsy

Exclusion Criteria:

* Excessive alcohol use (more than 20 g/day for women and 30g/day for men= >2 units alcohol/day for women and >3 units for men)
* Other liver diseases: Hepatitis B virus, Hepatitis C virus, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, Wilson's disease, Alpha 1 antitrypsin deficiency
* Secondary causes for steatosis: disorders of lipid metabolism, HCV Genotype 3, total parental nutrition, severe surgical weight loss, medications (amiodarone, tamoxifen, methotrexate, corticosteroids and HAART)
* Celiac disease
* pregnancy and breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-10-18 (Estimated); Study Completion 2024-10-18 (Estimated)

PRIMARY OUTCOMES:
Decrease in CAP (db/m) | 12 weeks
  The primary objective of this study is to determine the percentage decrease in hepatic steatosis at the end of week 12, measured by FibroScan® with CAP
Decrease in Liver Stiffness (kPa) | 12 weeks
  The primary objective of this study is to determine the percentage decrease in hepatic fibrosis at the end of week 12, measured by FibroScan® with E

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Banu Gungor, Prof, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa Hospital, Istanbul, Turkey (Türkiye)